CLINICAL TRIAL: NCT01305395
Title: Early Vs Late Sirolimus-Initiation Strategies To Prevent Cardiac Allograft Vasculopathy Related Events in Heart Transplant Recipients
Brief Title: Strategies To Prevent Cardiac Allograft Vasculopathy Related Events in Heart Transplant Recipients
Acronym: STOPCAV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due in part, to reduced transplant volume and enrollment has been difficult.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1007M85473
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Cardiac Allograft Vasculopathy in Heart Transplant
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Early Intervention Arm (Experimental): Initiate sirolimus within 6 months of heart transplant
  Interventions: Drug: Sirolimus
- Late Intervention Arm: Group 2A (Experimental): Initiate sirolimus after CAV is diagnosed by angiogram
  Interventions: Drug: Sirolimus
- Retrospective Arm: Angiogram group (Experimental): Start sirolimus after CAV diagnosed is by angiogram
  Interventions: Drug: Sirolimus
- Late Intervention Arm: Group 2B (Experimental): Start sirolimus after CAV is diagnosed by IVUS
  Interventions: Drug: Sirolimus
- Retrospective Arm: Intravascular Ultrasound (Experimental): Sirolimus after CAV is diagnosed by IVUS
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Will initiate sirolimus within 6 months of heart transplant
  Other Names: Rapamycin
  Arms: Early Intervention Arm
Drug: Sirolimus — Will start sirolimus after CAV has been diagnosed by angiogram
  Other Names: Rapamycin
  Arms: Late Intervention Arm: Group 2A
Drug: Sirolimus — Will start sirolimus after CAV has been diagnosed by intravascular ultrasound
  Other Names: Rapamycin
  Arms: Late Intervention Arm: Group 2B
Drug: Sirolimus — Will start sirolimus after they develop CAV by angiogram
  Other Names: Rapamycin
  Arms: Retrospective Arm: Angiogram group
Drug: Sirolimus — Will start sirolimus after CAV has been diagnosed by intravascular ultrasound
  Other Names: Rapamycin
  Arms: Retrospective Arm: Intravascular Ultrasound

SUMMARY:
1. Early initiation of sirolimus will prevent or delay the development of intimal thickening and subsequent graft failure.
2. Treatment guided by the development of cardiac allograft vasculopathy (CAV) on intravascular ultrasound (IVUS) will be more effective in delaying progression of CAV compared to treatment guided by angiography.
3. Prevention of the development and progression of intimal thickness on IVUS will prevent the development of heart failure, graft dysfunction, and cardiovascular death related to CAV.
4. Small artery elasticity predicts progression of cardiac allograft vasculopathy and is modified by sirolimus
5. Patients who have no progression of CAV will have favorable improvement in biomarkers and endothelial cells compared to patients who have progression of CAV

DETAILED DESCRIPTION:
Proliferation signal inhibitors (PSIs), sirolimus and everolimus, have been demonstrated to be effective immunosuppressants and delay the progression of cardiac allograft vasculopathy. To date, there are no prospective studies designed to evaluate the potential use of PSIs as a primary immunosuppressant in the prevention of cardiac allograft vasculopathy. The goals of our study are to compare primary vs. secondary preventive strategies and to evaluate the role of intravascular ultrasound compared to coronary angiogram in diagnosing CAV and preventing CAV-related events. The specific aims of the study are:

1. To evaluate the effect of primary vs. secondary initiation of sirolimus on the development of significant coronary artery (> 70% angiographic stenosis, Mean intimal thickness (MIT) 0.5mm or greater, IVUS calculated coronary cross sectional area of < 4mm2 / <6mm2 for mid LAD/Left Maim (LM), < 0.75 fractional flow reserve (FFR) lesion associated with a positive stress test), change in global left ventricle (LV) function, incidence of rejection episodes, and hospitalizations at 1, 2, 3, and 4 years.
2. To determine the effect of IVUS-guided initiation of sirolimus on short-term and long-term outcomes vs. angiogram-guided initiation of sirolimus
3. To determine whether prevention of progression of CAV diagnosed by IVUS prevents graft dysfunction or death related to CAV or heart failure.
4. To assess the correlation between peripheral small artery elasticity, peripheral biomarkers, and endothelial cells, and development of cardiac allograft vasculopathy in order to develop a strategy for determining risk of progression and monitoring treatment.

The study has a prospective and a retrospective arm

Prospective Arm Design: This is a prospective, randomized, partially-blinded pilot study. Randomization for the study will be done in 2 stages.

The first stage of randomization will randomize subjects to either the early or late initiation of sirolimus. At this stage of the randomization, subject will have a 30% chance of being in group 1 (early-initiation of sirolimus), and a 70% chance of being in group 2 (diagnostic-guided sirolimus group).

The second stage randomization will be done only on subjects in group 2 (diagnostic-guided sirolimus group) at the time of their first annual heart transplant review. At the time of their annual heart transplant review, subjects in group 2 will have a 50% chance of being in group 2A (CAV diagnosed by angiogram), and a 50% chance of being in group 2B (CAV diagnosed by intravascular ultrasound).

Group 1: Initiate sirolimus at 6 months after transplant

Group 2A: Initiate sirolimus after development of angiographic stenosis of >70% in a major epicardial vessel or >50% in the left main artery

Group 2B: Initiate sirolimus after development of maximal intimal thickness of 0.5 mm on intravascular ultrasound

Retrospective Arm

The main objective of this retrospective study is to compare a treatment strategy based on the diagnosis of CAV by intravascular ultrasound to a strategy guided by angiogram.

Design: This is a randomized, partially-blinded pilot study. Subjects will be randomized 1:1 to one of two groups. At the time of the randomization, the subject will have a 50% chance of being in group 1 (initiation of sirolimus when CAV is diagnosed by angiogram) and a 50% chance of being in group 2. (Initiation of sirolimus when CAV is diagnosed by IVUS)

Primary Endpoints for Prospective and Retrospective Arms

1. Change in maximal intimal thickness at 1, 2, 3 and 4 years
2. Combination of significant coronary artery disease (as described above), death, major rejection episodes, and decrease in global ejection function of more than 10% from baseline at 3 and 4years.

Secondary endpoints for Prospective and Retrospective Arms

1. Mean MIT at 1, 2, 3, and 4 years
2. Percent atheroma volume at 1,2,3 and 4 years
3. Death from CAV, death from any cause, myocardial infarction, need for PCI, number of hospitalizations, infection rates, evidence of restrictive physiology, arrhythmic event related to CAV or pulmonary hypertension at 4 years.
4. Change in small artery elasticity at 1, 2, 3, and 4 years
5. Change in endothelial progenitor cell count at 1 and 2 years
6. Change in biomarkers (see table) at 1 and 2 years

ELIGIBILITY:
Inclusion Criteria

For Prospective Arm:

* 18 years or older
* Successful orthotropic heart transplant within 6 months of enrollment

Inclusion Criteria

For Retrospective Arm:

* 18 years or older
* Successful orthotropic heart transplant within 6 months to 3 years of enrolment
* Less than moderate CAV by angiogram or IVUS

Exclusion Criteria

For Prospective Arm:

* Greater than minimal baseline coronary disease
* Chronic kidney disease with creatinine >2mg/dl
* Baseline (1 month) ejection fraction < 50%
* IV contrast allergy
* Rejection within 3 months of enrollment
* Sensitivity to sirolimus or its derivatives
* Prior sirolimus use

Exclusion Criteria

For Retrospective Arm:

* Significant baseline (one month) coronary artery disease (>50% in one or more vessels by angiogram or MIT >0.5 by IVUS)
* Chronic kidney disease with creatinine >2mg/dl
* Baseline (1 month) ejection fraction < 50%
* IV contrast allergy
* Rejection within 3 months prior to enrollment
* Sensitivity to sirolimus or its derivatives
* Prior sirolimus use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
1. Change in maximal intimal thickness | 1, 2, 3 and 4 years

SECONDARY OUTCOMES:
Mean maximal intima thickness | 1, 2, 3, and 4 years
Percent atheroma volume | 1,2,3 and 4 years
Death from CAV, death from any cause, myocardial infarction, need for percutaneous coronary intervention (PCI), number of hospitalizations, infection rates, evidence of restrictive physiology, arrhythmic event related to CAV or pulmonary hypertension | at 4 years.
Change in small artery elasticity | At 1, 2, 3, and 4 years
Change in endothelial progenitor cell count | At 1 and 2 years
Change in biomarkers | At 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Colvin-Adams, MD, MS, Principal Investigator — University of Minnesota
Locations (1):
- Cardiology Division, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Christie JD, Edwards LB, Aurora P, Dobbels F, Kirk R, Rahmel AO, Stehlik J, Taylor DO, Kucheryavaya AY, Hertz MI. The Registry of the International Society for Heart and Lung Transplantation: Twenty-sixth Official Adult Lung and Heart-Lung Transplantation Report-2009. J Heart Lung Transplant. 2009 Oct;28(10):1031-49. doi: 10.1016/j.healun.2009.08.004. No abstract available. PMID 19782285
- [Background] Rahmani M, Cruz RP, Granville DJ, McManus BM. Allograft vasculopathy versus atherosclerosis. Circ Res. 2006 Oct 13;99(8):801-15. doi: 10.1161/01.RES.0000246086.93555.f3. PMID 17038650
- [Background] Weis M, von Scheidt W. Cardiac allograft vasculopathy: a review. Circulation. 1997 Sep 16;96(6):2069-77. doi: 10.1161/01.cir.96.6.2069. PMID 9323100
- [Background] Johnson DE, Alderman EL, Schroeder JS, Gao SZ, Hunt S, DeCampli WM, Stinson E, Billingham M. Transplant coronary artery disease: histopathologic correlations with angiographic morphology. J Am Coll Cardiol. 1991 Feb;17(2):449-57. doi: 10.1016/s0735-1097(10)80114-7. PMID 1991903
- [Background] Rickenbacher PR, Pinto FJ, Chenzbraun A, Botas J, Lewis NP, Alderman EL, Valantine HA, Hunt SA, Schroeder JS, Popp RL, et al. Incidence and severity of transplant coronary artery disease early and up to 15 years after transplantation as detected by intravascular ultrasound. J Am Coll Cardiol. 1995 Jan;25(1):171-7. doi: 10.1016/0735-1097(94)00323-i. PMID 7798497
- [Background] Costello JM, Wax DF, Binns HJ, Backer CL, Mavroudis C, Pahl E. A comparison of intravascular ultrasound with coronary angiography for evaluation of transplant coronary disease in pediatric heart transplant recipients. J Heart Lung Transplant. 2003 Jan;22(1):44-9. doi: 10.1016/s1053-2498(02)00484-9. PMID 12531412
- [Background] Sharples LD, Jackson CH, Parameshwar J, Wallwork J, Large SR. Diagnostic accuracy of coronary angiography and risk factors for post-heart-transplant cardiac allograft vasculopathy. Transplantation. 2003 Aug 27;76(4):679-82. doi: 10.1097/01.TP.0000071200.37399.1D. PMID 12973108
- [Background] Kobashigawa JA, Tobis JM, Starling RC, Tuzcu EM, Smith AL, Valantine HA, Yeung AC, Mehra MR, Anzai H, Oeser BT, Abeywickrama KH, Murphy J, Cretin N. Multicenter intravascular ultrasound validation study among heart transplant recipients: outcomes after five years. J Am Coll Cardiol. 2005 May 3;45(9):1532-7. doi: 10.1016/j.jacc.2005.02.035. PMID 15862430
- [Background] Tuzcu EM, Kapadia SR, Sachar R, Ziada KM, Crowe TD, Feng J, Magyar WA, Hobbs RE, Starling RC, Young JB, McCarthy P, Nissen SE. Intravascular ultrasound evidence of angiographically silent progression in coronary atherosclerosis predicts long-term morbidity and mortality after cardiac transplantation. J Am Coll Cardiol. 2005 May 3;45(9):1538-42. doi: 10.1016/j.jacc.2004.12.076. PMID 15862431
- [Background] Mancini D, Pinney S, Burkhoff D, LaManca J, Itescu S, Burke E, Edwards N, Oz M, Marks AR. Use of rapamycin slows progression of cardiac transplantation vasculopathy. Circulation. 2003 Jul 8;108(1):48-53. doi: 10.1161/01.CIR.0000070421.38604.2B. Epub 2003 May 12. PMID 12742978
- [Background] Keogh A, Richardson M, Ruygrok P, Spratt P, Galbraith A, O'Driscoll G, Macdonald P, Esmore D, Muller D, Faddy S. Sirolimus in de novo heart transplant recipients reduces acute rejection and prevents coronary artery disease at 2 years: a randomized clinical trial. Circulation. 2004 Oct 26;110(17):2694-700. doi: 10.1161/01.CIR.0000136812.90177.94. Epub 2004 Jul 19. PMID 15262845
- [Background] Raichlin E, Bae JH, Khalpey Z, Edwards BS, Kremers WK, Clavell AL, Rodeheffer RJ, Frantz RP, Rihal C, Lerman A, Kushwaha SS. Conversion to sirolimus as primary immunosuppression attenuates the progression of allograft vasculopathy after cardiac transplantation. Circulation. 2007 Dec 4;116(23):2726-33. doi: 10.1161/CIRCULATIONAHA.107.692996. Epub 2007 Nov 19. PMID 18025531
- [Background] Raichlin E, Prasad A, Kremers WK, Edwards BS, Rihal CS, Lerman A, Kushwaha SS. Sirolimus as primary immunosuppression is associated with improved coronary vasomotor function compared with calcineurin inhibitors in stable cardiac transplant recipients. Eur Heart J. 2009 Jun;30(11):1356-63. doi: 10.1093/eurheartj/ehp123. Epub 2009 Apr 21. PMID 19383734